CLINICAL TRIAL: NCT07056231
Title: The Effect of Low Dose Caffeine on Serve Speed, Spike Speed, and Speed-Endurance in Elite Sitting Volleyball Players: A Randomized Double-Blind Crossover Study
Brief Title: Effect of Low-Dose Caffeine on Performance in Elite Sitting Volleyball Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ulaç Can YILDIRIM (Other)
Responsible Party: Sponsor-Investigator, Ulaç Can YILDIRIM, Assoc. Prof., Sinop University
Organization: Sinop University (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2025/91
Record Dates: First submitted 2025-06-21; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Caffeine; Physical Endurance; Muscle Strength; Paralympic Athletes
MeSH Terms: interventions — Caffeine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-Dose Caffeine Arm (Experimental): Participants receive a single oral dose of caffeine (3 mg/kg) during the first session and a placebo in the second session. There is a washout period of at least 48 hours between sessions.
  Interventions: Dietary Supplement: Caffeine; Dietary Supplement: Placebo
- Placebo Arm (Experimental): Participants receive a placebo during the first session and a single oral dose of caffeine (3 mg/kg) in the second session. There is a washout period of at least 48 hours between sessions.
  Interventions: Dietary Supplement: Caffeine; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Caffeine — A single oral dose of 3 mg of caffeine per kilogram of body weight form approximately 60 minutes before performance testing. Supplied by Oxford Vitality, ISO-certified.
Dietary Supplement: Placebo — polydextrose used as Placebo

SUMMARY:
Background: Sitting volleyball is a sport that relies primarily on upper body strength and anaerobic capacity. In critical in-game skills such as serve and spike, factors such as speed-endurance time and impact power play a decisive role in performance. There are limited studies in the literature examining the effects of low-dose caffeine consumption on these skills. The effects of ergogenic supplements in Paralympic sports have not been sufficiently investigated, and the potential benefits of caffeine on serve and spike performance in sitting volleyball players remain unclear. Purpose: The main purpose of this research was to determine the effects of low-dose caffeine (3 mg/kg) consumption on the serve speed, spike speed and Speed-Endurance performances of elite-level sitting volleyball players. Method: The study was designed using a randomized, double-blind, balanced, and crossover experimental design. 13 elite male athletes from the 2024 Paravolley European Champion Sitting Volleyball Men's National Team participated in the study. Participants were evaluated for serve speed, spike speed, and speed-endurance performances in both 3 mg/kg caffeine (CAF) and placebo (PLA) conditions.

DETAILED DESCRIPTION:
This study aimed to investigate the effects of low-dose caffeine ingestion on key performance parameters in elite-level sitting volleyball athletes. Sitting volleyball is a Paralympic sport that relies heavily on upper body explosive strength and short-term anaerobic power. While caffeine is a well-known ergogenic aid in able-bodied sports, its role in Paralympic contexts remains underexplored. Using a randomized, double-blind, placebo-controlled crossover design, the effects of 3 mg/kg caffeine consumption were assessed in 13 elite male sitting volleyball players. Each participant completed performance assessments under both caffeine and placebo conditions. The primary goal was to examine whether caffeine intake would enhance serve speed, spike speed, and repeated sprint ability. The study provides new insights into the acute ergogenic effects of caffeine in Paralympic team sport athletes, highlighting its selective benefit on explosive upper-body tasks such as serving.

ELIGIBILITY:
Inclusion Criteria:

* Male sitting volleyball players aged between 18 and 40
* Member of the 2024 National Sitting Volleyball Team
* At least 3 years of competitive playing experience
* No caffeine consumption 48 hours prior to testing
* Provided informed consent to participate

Exclusion Criteria:

* Known cardiovascular, neurological, or metabolic disorders
* Current use of medications that may affect caffeine metabolism
* Allergy or sensitivity to caffeine
* Use of performance-enhancing substances within the last month

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2025-03-05 (Actual); Primary Completion 2025-03-11 (Actual); Study Completion 2025-03-12 (Actual)

PRIMARY OUTCOMES:
Serve Speed | After 60 minutes ingestion of the supplement on test day (CAF and PLA)
  Serve speed will be assessed using a calibrated radar device to record peak velocity of each participant's volleyball serve.
Spike Speed | After 60 minutes ingestion of the supplement on test day (CAF and PLA)
  Maximum spike speed will be measured in kilometers per hour (km/h) using a radar gun during a standardized spike task conducted after supplementation in each condition.
Speed-Endurance | After 60 minutes ingestion of the supplement on test day (CAF and PLA)
  The number of maximal shuttle runs completed in a repeated sprint ability (RSA) test protocol will be recorded to assess speed-endurance capacity.

CONTACTS AND LOCATIONS:
Overall Officials: Ulas C Yildirim, Study Chair — sinop university faculty of sport sciences
Locations (1):
- Karamanoğlu Mehmetbey University, Karaman, Central, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Diedhiou AB, Erkan D, Guler M, Sar H, Karakulak I, Eyuboglu E, Gundem MC, Karayigit R, Tuncer SY, Yildirim UC. The effect of low dose caffeine powder supplementation on serve speed, spike speed, and speed-endurance in elite sitting volleyball players: a randomized double-blind crossover study. BMC Sports Sci Med Rehabil. 2025 Nov 6;17(1):320. doi: 10.1186/s13102-025-01408-8. PMID 41199325

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-06-28): https://cdn.clinicaltrials.gov/large-docs/31/NCT07056231/Prot_SAP_000.pdf